CLINICAL TRIAL: NCT05396001
Title: A Just-In-Time Adaptive Mobile Application Intervention To Reduce Sodium Intake And Blood Pressure In Hypertensive Patients: LowSalt4Life
Brief Title: LowSalt4Life: A Mobile Application to Reduce Sodium Intake And Blood Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Brahmajee K Nallamothu, Stevo Julius Research Professor of Cardiovascular Medicine and Professor of Internal Medicine, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HUM00210954; 1R61HL155498-01A1 (NIH)
Record Dates: First submitted 2022-05-24; First posted 2022-05-27 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Hypertension; Blood Pressure
Keywords: Dietary sodium
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants randomized to the App+JITAI will receive push notifications throughout the study, while those in the App alone group will not. The participants will not be told the group in which they are randomized, but they may know the group because of the number of push notifications.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LowSalt4Life (Active Comparator)
  Interventions: Behavioral: LowSalt4Life Application
- LowSalt4Life + just-in-time adaptive intervention (JITAI) (Experimental)
  Interventions: Behavioral: LowSalt4Life Application; Behavioral: Just-In-time Adaptive Intervention (JITAI)

INTERVENTIONS:
Behavioral: LowSalt4Life Application — LowSalt4Life is a dietary sodium intervention mobile application that promotes lower sodium intake.
Behavioral: Just-In-time Adaptive Intervention (JITAI) — LowSalt4Life is a dietary sodium application with a just-in-time adaptive intervention (JITAI) component enabled.
  Arms: LowSalt4Life + just-in-time adaptive intervention (JITAI)

SUMMARY:
This research is being done to learn if a smartphone app with and without a just in time adaptive intervention (JITAI) can help patients with hypertension manage their sodium intake and improve their blood pressure.

DETAILED DESCRIPTION:
The primary and secondary outcomes will be determined in months 1 & 2. Participants will continue for another 4 months and during that time data for exploratory measures will be collected.

During the first 2 months of the study, a micro-randomized trial (MRT) will be performed within the App+JITAI group (N=200). This MRT is designed to learn which push notification messages effectively prompt the user to interact with the appropriate content within the mobile application.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with essential hypertension (HTN) by a medical provider and are on stable doses of antihypertensive therapy for at least three months prior to enrollment as documented in the electronic health record (EHR) and confirmed by participant self-report.
2. A smartphone with a compatible Apple or Android operating system installed and able to download and use LowSalt4Life app including accepting all permissions and willing to allow the mobile applications to send push notifications
3. A valid email address
4. Fluent in spoken and written English

Exclusion Criteria:

1. Unstable symptoms or markedly elevated blood pressure (BP) at enrollment (defined as systolic BP>180 mmHg, diastolic BP>120 mmHg)
2. Contraindication to a sodium restriction diet
3. An estimated sodium intake less than 1,500mg per day
4. Known secondary causes of HTN (e.g., adrenal insufficiency, pheochromocytoma)
5. Estimated glomerular filtration rate (EGFR) <30 or end-stage renal disease on dialysis
6. Heart failure
7. Inability to use Withings devices (blood pressure cuff and scale) due to equipment limitations or contraindications
8. Currently pregnant or intent to become pregnant during the study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 410 (Actual)
Dates: Start 2022-08-15 (Actual); Primary Completion 2025-10-31 (Actual); Study Completion 2025-10-31 (Actual)

PRIMARY OUTCOMES:
Change in systolic blood pressure (SBP) | Baseline, 2 months
  SBP measured by a wireless home blood pressure monitor

SECONDARY OUTCOMES:
Change in weight over 2 months | Baseline, 2 months
  Weight measured using wireless scale
Change in estimated sodium intake | Baseline, 2 months
  As measured by the Block 2014 Food Frequency Questionnaire
Change in dietary nutrient intake | Baseline, 2 months
  As measured by the Block 2014 Food Frequency Questionnaire
Changes in blood pressure (BP) medications | Baseline, 2 months
  As measured by the electronic health record
Percent of participants at a goal blood pressure (BP) | 2 months
  Goal BPs are based on the American Heart Association blood pressure guidelines.

CONTACTS AND LOCATIONS:
Overall Officials: Brahmajee Nallamothu, Principal Investigator — University of Michigan
Locations (1):
- The University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
The aim is to prepare data for deposit into the National Heart, Lung, and Blood Institute (NHLBI) supported Biologic Specimen and Data Repositories Information Coordinating Center (BioLINCC).Unique research data be made available to the scientific community after the conclusion of a study. The de-identified analytic data will be prepared as SAS transport files or ASCII comma-delimited files with accompanying codebooks that describe the data and data structure. The redaction will employ best practices and will be consistent with National Heart, Lung, and Blood Institute data sharing policies.
Supporting Information: Study Protocol, ICF
Time Frame: Unique research data be made available to the scientific community after the conclusion of a study. No later than 3 years after the end of the study or 2 years after the main paper reporting the results of the trial, whichever comes first.
Access Criteria: The scientific community will have access to the data deposited into the National Heart, Lung, and Blood Institute (NHLBI) supported Biologic Specimen and Data Repositories Information Coordinating Center (BioLINCC). Researchers at institutions with a Federal Wide Assurance will be able to gain access to repository data by submitting a data access request in accordance with applicable policies.
URL: https://biolincc.nhlbi.nih.gov/

DOCUMENTS (1):
  • Informed Consent Form (2025-02-10): https://cdn.clinicaltrials.gov/large-docs/01/NCT05396001/ICF_000.pdf